CLINICAL TRIAL: NCT04543227
Title: The Impact of Ohio's Opioid Prescriptions Law on Opioid Use and Outcomes in Pediatric Patients
Brief Title: Opioid Laws and Pediatric Use
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Ohio Department of Public Safety (Unknown)
Responsible Party: Principal Investigator, Henry Xiang, Professor and Center Director, Nationwide Children's Hospital
Other Study IDs: STUDY00001192
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Burns; Knee Injuries; Opioid Use; Pain
Keywords: Burns; Knee Arthroscopy; Opioid; Pain; Chronic
MeSH Terms: conditions — Burns; Knee Injuries; Pain; Bronchiolitis Obliterans Syndrome | interventions — Aftercare

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Retrospective Burn Injuries: Pediatric patients treated at a large academic pediatric medical center for burn injuries between August 2015 - August 2019.
- Retrospective Knee Arthroscopy: Pediatric patients treated at a large academic pediatric medical center for a knee arthroscopy procedure between August 2015 - August 2019.
- Prospective Burn Injuries: Pediatric patients treated at a large academic pediatric medical center for burn injuries after July 2020.
  Interventions: Behavioral: Opioid Use 90-Days Post Treatment
- Prospective Knee Arthroscopy: Pediatric patients treated at a large academic pediatric medical center for a knee arthroscopy procedure after July 2020.
  Interventions: Behavioral: Opioid Use 90-Days Post Treatment

INTERVENTIONS:
Behavioral: Opioid Use 90-Days Post Treatment — Survey conducted 90-days post treatment to determine use of opioid medications in relation to burn or knee arthroscopy pain
  Groups: Prospective Burn Injuries; Prospective Knee Arthroscopy

SUMMARY:
The legitimate need for opioid medications for acute pain management in pediatric trauma patients is recognized, however, the high dose and duration of opioid drugs prescribed by medical providers has been associated with an increased risk of opioid abuse and chronic use by patients. The overarching goal of application is to assess opioid use and outcomes of pediatric patients treated for either burn injuries or knee arthroscopy procedures at a large academic pediatric medical center before and after Ohio opioid prescription rules for acute pain were implemented on August 21, 2017. Also, to evaluate patient use of opioids at 90-days post-treatment.

DETAILED DESCRIPTION:
This study has a prospective and retrospective component. Phase 1 involves a retrospective chart review will be performed among pediatric patients undergoing burn care or knee arthroscopy at our institution to determine a whether there was a reduction in prescribed opioid medications following the 2017 Ohio opioid prescription law. A 24-month pre-law period (August 1st, 2015, to August 31st, 2017) and 24-month post-law period (September 1st, 2017, to August 31st 2019) will be compared. This phase will include 300 patients (n=150 burn, n=150 knee arthroscopy) evenly divided between the pre-law and post-law periods.

Phase 2 involves a prospective patient telephone survey 90 days after burn care or knee arthroscopy procedure to assess the association of opioid prescribing, consumption and amount of left-over medications, and pain control status after 90 days. This phase will include 100 patients (n=50 burn, n=50 knee arthroscopy) recruited via convenience sampling.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients age 0-18 years (inclusive)
* treated at our institution for either a burn injury or knee arthroscopy procedure
* received at least one opioid prescription

Exclusion Criteria:

* patients age 19 years and above
* patients who did not receive any opioid medications
* patients undergoing knee arthroscopy with simultaneous anterior cruciate ligament (ACL) reconstruction
* families unable to to communicate in English

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients (age 0-18 years) treated at our institution for either a burn injury or knee arthroscopy procedure and received an opioid prescription.
Sampling Method: Non-Probability Sample
Enrollment: 980 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-11-16 (Actual)

PRIMARY OUTCOMES:
Change in opioid prescriptions | 2 years before and 2 years after Ohio opioid law
  Change in opioid medications prescribed pre-law and post-law (reported in morphine equivalent doses)
Long-term opioid use | 90 days post treatment
  Patients using opioid medications 90-days post treatment

SECONDARY OUTCOMES:
Comparison of opioid medications usage | 2 years before and 2 years after Ohio opioid law
  Comparison of opioid medications prescribed by injury type (burn and knee arthroscopy)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Xiang, MD, MPH, PhD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Armstrong M, Groner JI, Samora J, Olbrecht VA, Tram NK, Noffsinger D, Boyer EW, Xiang H. Impact of opioid law on prescriptions and satisfaction of pediatric burn and orthopedic patients: An epidemiologic study. PLoS One. 2023 Nov 16;18(11):e0294279. doi: 10.1371/journal.pone.0294279. eCollection 2023. PMID 37972014